CLINICAL TRIAL: NCT00303927
Title: Thymidylate Synthase (TS) Genotype-Directed Phase II Trial of Oral Capecitabine for 2-Line Treatment of Advanced Pancreatic Cancer
Brief Title: Capecitabine as Second-Line Therapy in Treating Patients With Stage IV Pancreatic Cancer Who Have the Thymidylate Synthase Gene
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Wells Messersmith, Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000462118; P30CA006973 (NIH); JHOC-J0560; JHOC-NA_00000937
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2010-03

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine

INTERVENTIONS:
Drug: capecitabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well capecitabine works as second-line therapy in treating patients with stage IV pancreatic cancer who have the thymidylate synthase gene.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Characterize the 6-month survival of patients with stage IV pancreatic cancer (progressing after at least 1 prior gemcitabine-containing chemotherapy regimen) who carry the double tandem repeat (S/S) variant of the thymidylate synthase (TS) gene enhancer region (TSER) treated with capecitabine.
* Characterize toxicity of capecitabine in patients with stage IV pancreatic cancer who carry the S/S variant of the TSER.

Secondary

* Explore the association between capecitabine exposure at steady-state, allelic variants in candidate genes (carboxylesterase 1, carboxylesterase 2, cytidine deaminase, thymidine phosphorylase [TP], dihydropyrimidine dehydrogenase [DPD], methylenetetrahydrofolate reductase) and drug response (toxicity and efficacy) in this patient population.
* Determine the relationship between expression of TS, TP, and DPD in tumor tissues and the response to capecitabine in this patient population.
* Analyze response rate to capecitabine, based on the presence of homozygous S/S variant of the TSER.

OUTLINE: This is an open-label, multicenter study.

Patients receive oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 65 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed pancreatic cancer

  * Stage IV disease
* Measurable disease (≥ 1 cm or > 10 mm lesion(s) by spiral CT scan)
* Disease progression after ≥ 1 gemcitabine-based treatment regimen for advanced/metastatic disease
* Patient carries the double tandem repeat (S/S) variant of the thymidylate synthase gene enhancer region (TSER)
* No active CNS metastases (indicated by clinical symptoms, cerebral edema, steroid requirement, or progressive growth)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* AST/ALT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if attributable to liver metastases)
* Total bilirubin ≤ 1.5 times ULN
* Creatinine normal OR creatinine clearance > 50 mL/min
* Fertile patients must use effective contraception during and for 30 days after completion of study treatment
* Not pregnant or nursing
* Negative pregnancy test
* Asymptomatic HIV infection allowed
* No recent or ongoing clinically significant gastrointestinal disorder (e.g., malabsorption, bleeding, inflammation, emesis, or diarrhea > grade 1)
* Able to swallow capecitabine tablets
* No known hypersensitivity to fluorouracil
* No dihydropyrimidine dehydrogenase (DPD) deficiency
* No clinically significant cardiac disease (e.g., congestive heart failure, symptomatic coronary artery disease, or cardiac arrhythmias not well controlled with medication)
* No myocardial infarction within the past 6 months
* No serious, uncontrolled, concurrent infection(s)
* No prior unanticipated severe reaction to fluoropyrimidine therapy
* No other malignancy within the past 5 years except cured nonmelanoma skin cancer or treated carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy
* No prior capecitabine except in the adjuvant setting
* At least 3 weeks since prior radiotherapy or major surgery
* At least 4 weeks since prior participation in any investigational drug study
* At least 4 weeks since prior sorivudine or brivudine
* No concurrent sorivudine or brivudine
* No concurrent cimetidine or azidothymidine (AZT)
* Concurrent radiotherapy for bone pain allowed to a limited field provided ≥ 1 indicator lesion remains outside of the field
* No other concurrent chemotherapy or immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2005-12; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Survival at 6-months
Toxicity

SECONDARY OUTCOMES:
Association between capecitabine exposure at steady-state, allelic variants in candidate genes, and drug response
Relationship between expression of TS, TP and DPD in tumor tissues and response
Response rate

CONTACTS AND LOCATIONS:
Overall Officials: Wells Messersmith, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States
- Hospital Universitario 12 de Octubre, Madrid, Spain